CLINICAL TRIAL: NCT01392989
Title: Post Transplant Infusion of Allogeneic Cytokine Induced Killer Cells as Consolidative Therapy After Non-Myeloablative Allogeneic Transplantation in Patients With Myelodysplasia or Myeloproliferative Disorders
Brief Title: Post T-plant Infusion of Allogeneic Cytokine Induced Killer (CIK) Cells as Consolidative Therapy in Myelodysplastic Syndromes/Myeloproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Everett Meyer (Other)
Responsible Party: Sponsor-Investigator, Everett Meyer, Assistant Professor-Med, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18127; SU-04202010-5724 (Other: Stanford University); BMT217 (Other: OnCore)
Record Dates: First submitted 2011-06-21; First posted 2011-07-13 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Neural Tube Defects; Anemia; Leukemia, Myeloid; Bone Marrow Transplant Failure; Myelodysplastic Syndromes (MDS); Myeloproliferative Disorders
MeSH Terms: conditions — Neural Tube Defects; Anemia; Leukemia, Myeloid; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Cyclosporine; Mycophenolic Acid; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic Cytokine-induced Killer Cells (CIK) (Experimental): Target dose of ≥ 5 x 10e6 CD34+ cells/kg of recipient body weight plus an additional 2 x10e9 mononuclear cells.
  Interventions: Drug: CIK cells; Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Drug: Thymoglobulin; Radiation: Total Lymphoid Irradiation (TLI)

INTERVENTIONS:
Drug: CIK cells — Standard of care
  Other Names: Cytokine-induced Killer Cells
Drug: Cyclosporine — 5 mg/kg, po
  Other Names: cyclosporin; cyclosporin A
Drug: Mycophenolate Mofetil — 15 mg/kg, oral
  Other Names: MMF; CellCept
Drug: Thymoglobulin — 7.5 mg/kg, IV
  Other Names: Anti-thymocyte globulin; ATG
Radiation: Total Lymphoid Irradiation (TLI)

SUMMARY:
Allogeneic stem cell transplantation (transplant of blood cells from another individual) is a treatment option for patients with myelodysplasia or myeloproliferative Disorders. During the course of this study, it will be evaluated whether a particular type of blood cell, called a cytokine-induced killer (CIK) cell, may add benefit to allogeneic stem cell transplantation. CIK cells are present in small quantities in the bloodstream but their numbers can be expanded after a brief period of nurturing in a laboratory.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the rate of conversion to FDC following infusion of allogeneic CIK cells among patients with MDS, therapy-related myeloid neoplasms, or MPD who receive non myeloablative preparative regimen of TLI / ATG followed by allogeneic HCT and consolidation with allogeneic CIK cells.

Secondary Objectives:

* To determine the 2 year overall survival (OS) and event free survival (EFS)
* To determine the incidence of acute GVHD following infusion of allogeneic CIK cells
* To assess the pre-transplant expression of NKG2D ligands in patients' bone marrow aspirates.

ELIGIBILITY:
INCLUSION CRITERIA, RECIPIENT WITH MYELODYSPLASTIC SYNDROME (MDS)

* Diagnosis of MDS classifiable by the World Health Organization (WHO) on the basis of:

  * Refractory anemia
  * Refractory anemia with excess blasts-1
  * Refractory anemia with excess blasts-2
  * Refractory cytopenia with multi-lineage dysplasia
  * Refractory cytopenia with multi-lineage dysplasia and ringed sideroblasts
  * Chronic myelomonocytic leukemia (CMML)
  * MDS transformed to acute leukemia
  * MDS-unclassified
* Participants with advanced MDS must have < 10% marrow blasts prior to receiving conditioning with TLI/ATG, documented by marrow examination within 1 month prior.
* Participants with evolution to acute leukemia (AML) must be in a morphologic leukemia free-state (MLFS) with blasts < 5%

INCLUSION CRITERIA, RECIPIENT WITH MYELOPROLIFERATIVE DISORDER (MPD)

* Diagnosis of MPD on the basis of:

  * Idiopathic myelofibrosis
  * Polycythemia vera
  * Essential thrombocythemia
  * Chronic myelomonocytic leukemia (CML)
  * CML, Philadelphia chromosome-negative
  * Chronic neutrophilic leukemia
  * Chronic eosinophilic leukemia
  * Hypereosinophilic cyndrome
  * Systemic mastocytosis
* < 10% marrow blasts prior to receiving conditioning with TLI/ATG, documented by marrow examination within 1 month prior.
* Participants with evolution to acute leukemia (AML) must be in a morphologic leukemia free-state (MLFS) with blasts < 5%. Presence of residual dysplastic features following cytoreductive therapy is acceptable.

INCLUSION CRITERIA, RECIPIENT WITH THERAPY-RELATED MYELOID NEOPLASM (t MDS)

* < 10% marrow blasts prior to receiving conditioning with TLI/ATG, documented by marrow examination within 1 month prior.
* Morphologic leukemia free-state with blasts < 5 %.
* Age > 50 years, or < 50 years of age but at high-risk for regimen-related toxicity associated with conventional myeloablative transplants due to pre-existing medical conditions or prior therapy
* Availability of a fully HLA-matched or single antigen/allele mismatched sibling or unrelated donor
* Prior malignancy diagnosed > 5 years ago without evidence of disease, or < 5 years ago with life expectancy of > 5 years are eligible (prior malignancy is not a requirement)

INCLUSION CRITERIA, DONOR

* Donors must be HLA-matched or one allele mismatched.
* Donor age < 75 (EXCEPTION by Principal Investigator discretion)
* Must consent to PBSC mobilization with G-CSF; apheresis; and collection and donation of plasma
* Donor must consent to placement of a central venous catheter in the event that peripheral venous access is limited.

EXCLUSION CRITERIA, RECIPIENT

Any of the following:

* Uncontrolled CNS involvement with disease
* Pregnant
* Cardiac function: ejection fraction (EF) < 35% or uncontrolled cardiac failure
* Diffusing capacity of the lungs for carbon monoxide (DLCO) < 40% predicted
* Bilirubin > 3 mg/dL
* Aspartate aminotransferase (AST) > 3x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 3x ULN
* Estimated creatinine clearance < 50 mL/min
* Karnofsky performance score (KPS) < 70%
* Documented fungal disease that is progressive despite treatment
* HIV-positive

EXCLUSION CRITERIA, DONOR

Any of the following:

* Identical twin to recipient
* Pregnant or lactating
* Prior malignancy within the preceding 5 years (EXCEPTION: non-melanoma skin cancers)
* HIV seropositivity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06-07 (Actual); Study Completion 2017-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Meyer, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narayan R, Benjamin JE, Shah O, Tian L, Tate K, Armstrong R, Xie BJ, Lowsky R, Laport G, Negrin RS, Meyer EH. Donor-Derived Cytokine-Induced Killer Cell Infusion as Consolidation after Nonmyeloablative Allogeneic Transplantation for Myeloid Neoplasms. Biol Blood Marrow Transplant. 2019 Jul;25(7):1293-1303. doi: 10.1016/j.bbmt.2019.03.027. Epub 2019 Apr 3. PMID 30951840

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic Cytokine Induced Killer Cells (CIK): Target dose of ≥ 5 x 106 CD34+ cells/kg of recipient body weight plus an additional 2 x109 mononuclear cells.
  CIK cells: Standard of care
  Cyclosporine: 5 mg/kg, po
  Mycophenolate Mofetil: 15 mg/kg, oral
  Thymoglobulin: 7.5 mg/kg, IV
Period: Total Lymphoid Irradiation (TLI)
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Started | 44
Completed | 44
Not Completed | 0
Period: CIK Cell Infusion
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Full Donor Chimerism (FDC)
Description: Proportion of patients achieving full donor T-cell chimerism (FDC) by on or before Day 90 post non-myeloablative allogeneic transplant with allogeneic cytokine-induced killer (CIK) cells will be determined. FDC is defined as the attainment of >95% donor type CD3+ cells. The outcome will be reported as number of participants who achieved full donor chimerism, a number without dispersion.
Time Frame: 90 days
Population: Cytokine-induced killer (CIK) cells were infused in a subset of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 31
Participants | 6

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is an expression of the number of participants that remain alive 2 years after cytokine-induced killer (CIK) infusion. The outcome will be reported as the number of participants alive 2 years after CIK infusion, a number without dispersion.
Time Frame: 2 years
Population: Cytokine-induced killer (CIK) cells were infused in a subset of participants. Participants that did not receive CIK cells were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 31
Participants | 16

3. Secondary Outcome: Event-free Survival (EFS) Rate
Description: Event-free Survival (EFS) rate will be assessed on all enrolled participants and is defined as the duration of time after cytokine-induced killer (CIK) cell infusion that the participants remain alive with experiencing relapse, Grade 3 to 4 acute graft vs host disease (aGVHD), or death. The outcome will be reported as the number of participants, stratified by receipt of CIK cells, that did not experience a specified event, a number without dispersion.
Time Frame: 2 years
Population: All participants are reported. Cytokine-induced killer (CIK) cells were infused in a subset of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 44
Participants
  CIK-infused participants: number analyzed (Participants) | 31
  CIK-infused participants | 14
  Non-CIK-infused participants: number analyzed (Participants) | 13
  Non-CIK-infused participants | 4

4. Secondary Outcome: Number of Participants That Experience Grade 2 to 4 aGvHD Within 100 Days and 1 Year
Description: Acute graft vs host disease (aGvHD) Grade 2 to 4 was staged & graded using modified Keystone criteria, as below. The outcome is reported as the number of participants that experience Grade 2 to 4 aGvHD within 100 days and 1 year.
  * Stage 1: Skin: rash < 25% of skin. Liver: bilirubin 2 to 3 mg/dL. Gut: diarrhea 500 to 1000 mL/day or persistent nausea with positive biopsy for GvHD
  * Stage 2: Skin: rash 25 to 50% of skin. Liver: bilirubin 3 to 6 mg/dL. Gut: diarrhea 1000 to 1500 mL/day.
  * Stage 3: Skin: rash > 50% of skin. Liver: bilirubin 6 to 15 mg/dL. Gut: diarrhea > 1500 mL/day.
  * Stage 4: Skin: generalized erythroderma with bulla formation. Liver: bilirubin > 15 mg/dL. Gut: severe abdominal pain with or without ileus Grade of aGvHD was determined as follows.
  * Grade 1: Stage 1-2 Skin + No Liver stage + No Gut stage
  * Grade 2: Stage 3 Skin OR Stage 1 Liver or Stage 1 Gut
  * Grade 3: No Skin stage + Stage 2 to 3 Liver Stage 2 to 4 Gut
  * Grade 4: Stage 4 Skin + or Stage 2
Time Frame: 1 year
Population: Cytokine-induced killer (CIK) cells were infused in a subset of participants. Results are reported for both subsets and collectively, at 2 time points.
Measure: Count of Participants; unit: Participants
Groups:
- Allogeneic Cytokine Induced Killer Cells (CIK): Target dose of ≥ 5 x 10e6 CD34+ cells/kg of recipient body weight plus an additional 2 x10e9 mononuclear cells.
  CIK cells: Standard of care
  Cyclosporine: 5 mg/kg, po
  Mycophenolate Mofetil: 15 mg/kg, oral
  Thymoglobulin: 7.5 mg/kg, IV
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 44
Participants
  All participants within 100 days | 9
  All participants within 1 year | 11
  CIK-infused participants within 100 days: number analyzed (Participants) | 31
  CIK-infused participants within 100 days | 3
  CIK-infused participants within 1 year: number analyzed (Participants) | 31
  CIK-infused participants within 1 year | 5
  Non-CIK-infused participants within 100 days: number analyzed (Participants) | 13
  Non-CIK-infused participants within 100 days | 6
  Non-CIK-infused participants within 1 year: number analyzed (Participants) | 13
  Non-CIK-infused participants within 1 year | 6

5. Secondary Outcome: Pre-transplant Expression of Natural-killer Group 2, Member D (NKG2D) Ligands
Description: Pre-transplant expression of natural-killer group 2, member D (NKG2D) ligands MIC A, MIC B, and the UL16 binding proteins (ULBPs) will be assessed in participants' bone marrow aspirates. The outcomes is expressed as the number of participants whose expression level for each ligand was elevated compared to background, represented by the known levels for individual without cancer.
Time Frame: Pre-transplant
Population: Insufficient tumor sample materials from the pre-transplant diagnostic bone marrow aspirate was available for the research analysis. No analysis was conducted.
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Allogeneic Cytokine Induced Killer Cells (CIK)
All-Cause Mortality (participants affected / at risk) | 24/44
Serious Adverse Events (participants affected / at risk) | 27/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Cytokine Induced Killer Cells (CIK) (N=44)
Fever (General disorders) | 1 (1)
Infections and infestations -Other, bacteremia (Infections and infestations) | 1 (1)
Death NOS (General disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, GvHD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Aspiration (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal and urinary disorders -Other, Renal failure (Renal and urinary disorders) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Cytokine Induced Killer Cells (CIK) (N=44)
Serum sickness (Immune system disorders) | 13 (16)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, cardiac bigeminy (Cardiac disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (6)
Dizziness (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Fever (General disorders) | 9 (11)
Non-cardiac chest pain (General disorders) | 1 (1)
General Disorders Other - Peripheral Edema (General disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders -Other, Diverticulitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Infections and infestations - Other , Catheter Infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Viremia (Infections and infestations) | 2 (2)
Infections and infestations - Other, Coronavirus (Infections and infestations) | 1 (1)
Platelet Count decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Weight Gain (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders -Other, Dysuria (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders Other, cutaneous eruptions (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders Other, Rash (Skin and subcutaneous tissue disorders) | 5 (8)
Hypertension (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders - Other, DVT (Vascular disorders) | 1 (1)
Psychiatric disorders - Other, altered mental status (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No